CLINICAL TRIAL: NCT05613270
Title: A Prospective Pilot Study to Explore Performance and Efficacy of 18F-FES PET/CT in ER-positive Breast Cancer Patients
Brief Title: Characterizing Breast Cancer With 18F-FES PET/CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-FES-BC-1
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FES PET/CT (Experimental): Inject 18F-FES and then perform PET/CT scan.
  Interventions: Diagnostic Test: 18F-FES PET/CT scan

INTERVENTIONS:
Diagnostic Test: 18F-FES PET/CT scan — Patients with suspected metastatic ER-positive breast cancer underwent 18F-FES PET/CT after an injection of 185-222 MBq (5-6 mCi) 18F-FES to image lesions of metastatic breast cancer.

SUMMARY:
18F-fluoroestradiol (FES) is radioactive labeled estradiol, developed for in vivo visualization of estrogen receptor (ER) using positron emission tomography (PET). In this prospective study, 18F-FES PET/CT will be used to evaluate ER activity of metastatic disease and their potential sensitivity to endocrine therapy in ER-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed metastatic ER-positive breast cancer;
* 18F-FDG PET/CT within two weeks;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 18F-FES in BC | through study completion, an average of 1 year
  The max standard uptake value (SUVmax) was measured in the breast cancer lesions on 18F-FES PET/CT.
Lesions detected by 18F-FES PET/CT | through study completion, an average of 1 year
  The number of target lesions was calculated by 18F-FES PET/CT.
Compared with 18F-FDG PET/CT | through study completion, an average of 1 year
  The number of lesions detected by 18F-FES PET/CT was compared with 18F-FDG PET/CT.

SECONDARY OUTCOMES:
Overall survival | 3 years
  Evaluate overall survival (OS) in patients receiving regimens containing endocrine therapy

CONTACTS AND LOCATIONS:
Overall Officials: Li Huo, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China